CLINICAL TRIAL: NCT04920929
Title: A Prospective, Randomized, PICC Asymptomatic Thrombosis Study: A Pilot Study
Brief Title: PICC Asymptomatic Thrombosis Study: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment too low, not meeting objectives
Sponsor: Access Vascular Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLIN 20-002
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Peripheral ICC

STUDY DESIGN:
Intervention Model Description: Randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hydrophilic BioMaterial (Active Comparator): Hydrophilic BioMaterial- HydroPICC
  Interventions: Device: Hydrophilic Biomaterial
- Thermoplastic Polyurethane (Active Comparator): TPU- 4 French Single Lumen PowerPICC
  Interventions: Device: Thermoplastic Polyurethane

INTERVENTIONS:
Device: Hydrophilic Biomaterial — PICC made out of a Hydrophilic Biomaterial
  Other Names: HydroPICC
  Arms: Hydrophilic BioMaterial
Device: Thermoplastic Polyurethane — PICC made out of a thermoplastic polyurethane material
  Other Names: PowerPICC
  Arms: Thermoplastic Polyurethane

SUMMARY:
The study purpose is to perform a preliminary, comparative evaluation of the Hydrophilic Biomaterial technology to confirm the performance of the catheter, by using UltraSound technology in-vivo.

DETAILED DESCRIPTION:
This study will compare two different materials to evaluate asymptomatic thrombosis using ultrasound technology.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is indicated for a medically necessary PICC for therapeutic delivery medication
2. Patient is eligible to receive a single lumen PICC
3. Patient is an adult who is prescribed a PICC line
4. Patient's expected duration of treatment requiring a PICC for a minimum of 16 days post device implantation
5. Patient understands and is willing to comply with all study requirements and has voluntarily signed the Informed Consent Form (ICF).

Exclusion Criteria:

1. Is pregnant, lactating, or is planning to become pregnant during the time of the study
2. Has been previously enrolled in this post market clinical evaluation, or is participating in another clinical study that is contraindicative to the treatment or outcomes of this investigation
3. Venous thrombosis in any portion of the vein to be catheterized
4. Conditions that impede venous return from the extremity such as paralysis or lymphedema after mastectomy
5. Orthopedic or neurological conditions affecting the extremity
6. Anticipation or presence of dialysis grafts or other intraluminal devices, including pacemakers, within a month of patient enrollment start
7. Patients who are on anticoagulation therapy prior to the study (10-14 days). Note: (If patients are placed on anticoagulation (low dose) therapy while hospitalized, these patients are allowed.)
8. Patient has relinquished control of care to a guardian and/or facility
9. Patient has any significant medical or physical condition that, in the opinion of the PI, would make the subject unsuitable for participation in the post market clinical evaluation
10. Inability to complete the protocol in the opinion of the clinical staff due to safety or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, MD, Principal Investigator — Beaumont Hospital
Locations (1):
- Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrophilic BioMaterial | Thermoplastic Polyurethane
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated due to enrollment difficulties and no analysis was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrophilic BioMaterial | Thermoplastic Polyurethane | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (14.24) | 63.3 (2.28) | 63.6 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Asymptomatic Thrombosis Rate
Description: Rate of asymptomatic thrombosis measured using ultrasound technology for each group
Time Frame: 7 days post insertion
Population: number of subjects with asymptomatic thrombosis measured at Day 7 post insertion using ultrasound technology
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrophilic BioMaterial | Thermoplastic Polyurethane
Number analyzed (Participants) | 3 | 4
Participants | 2 | 1

2. Secondary Outcome: Symptomatic Thrombosis Rate
Description: Rate of symptomatic thrombosis measured using ultrasound technology
Time Frame: 14 days post insertion
Population: number of subjects with symptomatic thrombosis measured using ultrasound technology at day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrophilic BioMaterial | Thermoplastic Polyurethane
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

3. Secondary Outcome: Symptomatic Thrombosis Rate
Description: Rate of symptomatic thrombosis measured using ultrasound technology
Time Frame: 7 days post insertion
Population: number of subjects with symptomatic thrombosis measured with ultrasound technology at day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrophilic BioMaterial | Thermoplastic Polyurethane
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 3 Months
Arm/Group | Hydrophilic BioMaterial | Thermoplastic Polyurethane
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrophilic BioMaterial (N=3) | Thermoplastic Polyurethane (N=4)
superficial venous thrombosis of arm (Vascular disorders) | 2 (2) | 1 (1)
left lower quadrant pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
lung Nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
deep venous thrombosis arm (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT04920929/Prot_SAP_000.pdf